CLINICAL TRIAL: NCT01206296
Title: A Phase 2 Study of Adjuvant Intraperitoneal Gemcitabine for Resectable Pancreatic Adenocarcinoma
Brief Title: Adjuvant Intraperitoneal Gemcitabine for Resectable Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study suspended
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCI 2009-455
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Adjuvant; Intraperitoneal; Gemcitabine; Pancreas; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraperitoneal Gemcitabine (Experimental): Intraperitoneal Gemcitabine
  Interventions: Drug: Intraperitoneal Gemcitabine

INTERVENTIONS:
Drug: Intraperitoneal Gemcitabine — Standard pancreatic resection followed by heated intraoperative intraperitoneal gemcitabine 1000 mg/m2
  Adjuvant intraperitoneal gemcitabine treatments (days 1, 8 and 15 of each 4-week cycle) for 6 cycles

SUMMARY:
This is a phase II study evaluating the use of intraperitoneal gemcitabine given intraoperatively and as adjuvant therapy for patients with resectable pancreas cancer.

The primary objective of this study is to evaluate the overall safety of intraperitoneal gemcitabine given intraoperatively and postoperatively for adjuvant treatment of resectable pancreatic adenocarcinoma.

The secondary objectives are to evaluate the efficacy of this treatment regimen as reflected in overall survival at 2-years, to study the patterns of disease recurrence following this treatment, to study the pharmacology of intraperitoneal gemcitabine and to study changes in peritoneal cytology with pancreatic cancer resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the pancreas or periampullary cancer (duodenum, ampulla of Vater or distal common bile duct).
* Patients without a histologically confirmed diagnosis prior to surgical exploration, will have intraoperative frozen section to confirm the diagnosis prior to the administration of intraoperative intraperitoneal gemcitabine.
* Patients must undergo adequate preoperative imaging evaluation to determine resectability including contrast enhanced CT scan or MRI with or without endoscopic ultrasound
* Patients must have a complete surgical resection to grossly negative margins. The margins will be assessed in a routine fashion: the surgeon will decide on the level of transection based on visual inspection making sure that the visible/palpable tumor is removed with a negative margin. The specimen will be assessed for pancreatic duct and bile duct margin by intraoperative frozen section and an attempt will be made to have microscopically negative margins in all cases.
* Patients who have not received chemotherapy for the treatment of their pancreatic cancer prior to surgery scheduled at the Washington Hospital Center may be included in the protocol.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of gemcitabine in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 2 combination trials.
* Life expectancy of greater than 6 months
* ECOG (Eastern Cooperative Oncology Group) performance status <2
* Patients must have normal organ and marrow function as defined below:
* leukocytes >3,000/mcL
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* total bilirubin within normal institutional limits or compatible with preoperative biliary obstruction caused by the tumor
* AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal or compatible with preoperative biliary obstruction caused by the tumor
* creatinine within normal institutional limits OR
* creatinine clearance >45 mL/min
* The effects of gemcitabine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to avoid pregnancy prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had radiotherapy or chemotherapy for their pancreatic cancer
* Patients receiving any other investigational agents.
* Patients with metastatic disease in the liver or other distant sites, intraabdominal lymph nodes beyond regional draining lymph nodes or with malignant ascites
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because gemcitabine is an antimetabolite (pyrimidine analog) with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with gemcitabine, breastfeeding should be discontinued if the mother is treated with gemcitabine. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with gemcitabine. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lana Bijelic, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- See also: Washington Hospital Center — https://www.medstarwashington.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraperitoneal Gemcitabine: Intraperitoneal Gemcitabine
  Intraperitoneal Gemcitabine: Standard pancreatic resection followed by heated intraoperative intraperitoneal gemcitabine 1000 mg/m2
  Adjuvant intraperitoneal gemcitabine treatments (days 1, 8 and 15 of each 4-week cycle) for 6 cycles
Period: Overall Study
Arm/Group | Intraperitoneal Gemcitabine
Started (The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. Additional efforts were made to obtain study data via publications, IRB and RedCap systems. No study data are available.) | 0
Completed (The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. Additional efforts were made to obtain study data via publications, IRB and RedCap systems. No study data are available.) | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful.
  Additional efforts were made to obtain study data via publications, IRB and RedCap systems.
  No study data are available.
Arm/Group | Intraperitoneal Gemcitabine
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Grade III and IV Complications
Description: Incidence of grade III and IV complications related to intraopertaive intraperitoneal gemcitabine occurring during hospitalization or within 30 days of surgery, whichever is longer
Time Frame: Occurring during hospitalization or within 30 days of surgery, whichever is longer
Population: as for baseline characteristics
Arm/Group | Intraperitoneal Gemcitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: N/A - The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. Additional efforts were made to obtain study data via publications, IRB and RedCap systems. No study data are available.
Description: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful.
  Additional efforts were made to obtain study data via publications, IRB and RedCap systems.
  No study data are available.
Arm/Group | Intraperitoneal Gemcitabine
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes